CLINICAL TRIAL: NCT04311060
Title: Genetic and Molecular Characteristics of Mexican Adults With Acute Myeloid Leukemia: a Prospective Multicenter Study
Brief Title: Genetic and Molecular Characteristics of Mexican Adults With Acute Myeloid Leukemia: a Prospective Multicentric Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mexican Agrupation for Hematology Study (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Instituto Nacional de Cancerologia de Mexico (Other); Centro Medico Nacional Siglo XXI IMSS (Other); Hospital General de México Dr. Eduardo Liceaga (Other Government); Hospital Regional de Alta Especialidad del Bajio (Other); Instituto Mexicano del Seguro Social (Other Government); Hospital Universitario Dr. Jose E. Gonzalez (Other); Hospital Regional de Alta Especialidad de Ciudad Victoria Bicentenario 2010 (Other); Hospital Juarez de Mexico (Other Government); Hospital Regional de Alta especialidad de Ixtapaluca (Other)
Responsible Party: Sponsor
Other Study IDs: HEM-3094-19-25-1
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Bone marrow samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Molecular panel — * Detection of CBF rearrangements using PCR: CBFB-MYH11 [inv(16)(p13;q22), isoforms A, E and D; AML-ETO (RUNX1-RUNX1T1) (t8;21)(q22;q22).
  * NGS panel to detect classic mutations in: FLT3-ITD and TKD, NPM1, CEBPA, RUNX1, TP53, ASXL1, IDH1, IDH2 and KIT

SUMMARY:
Newly diagnosed adults patients with Acute Myeloid Leukemia will be assessed as traditionally by the treating institution using classic clinical, demographic and cytogenetic variables. Complementary molecular tests will be performed in the patients included in the study using PCR to detect classic CBF (Core Binding Factor) rearrangements: CBFB-MYH11 [inv(16)(p13;q22), isoforms A, E and D; AML-ETO (RUNX1-RUNX1T1) (t8;21)(q22;q22). NGS (Next Generation Sequencing) to detect mutations in: FLT3-ITD and TKD, NPM1, CEBPA, RUNX1, TP53, ASXL1, IDH1, IDH2 and KIT

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML
* Over 15 years of age
* Flow cytometry confirmation
* Candidate for treatment (intensive or not intensive)

Exclusion Criteria:

* Acute Promyelocytic Leukemia
* Mixed phenotype leukemias
* Isolated myeloid sarcoma
* Blastic plasmacytoid dendritic cell neoplasm

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mexican adults with newly diagnosed AML who are candidates for treatment (intensive or not intensive)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-22 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 year

CONTACTS AND LOCATIONS:
Locations (10):
- Mexico (10):
  - Hospital Regional de Alta Especialidad Ixtapaluca, Ixtapaluca, Edo Mex
  - Hospital Regional de Alta Especialidad Bajío, León, Guanajuato
  - Hospital Universitario, Monterrey, Nuevo León
  - Imss Umae 25, Monterrey, Nuevo León
  - Hospital Regional de Alta Especialidad Ciudad Victoria, Ciudad Victoria, Tamaulipas
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City
  - Centro Médico Naciona Siglo XXI IMSS, Mexico City
  - Hospital General de México, Mexico City
  - Hospital Juarez de México, Mexico City
  - Instituto Nacional de Cancerlogía, Mexico City

IPD SHARING:
Plan to Share IPD: No